CLINICAL TRIAL: NCT05871957
Title: Adjuvant Therapeutic Effect of Vitamin D on Hashimoto's Thyroiditis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: YXLL-KY-2021(041)
Record Dates: First submitted 2022-10-15; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Hashimoto Thyroiditis
MeSH Terms: conditions — Hashimoto Disease | interventions — Vitamin D

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Serum vitamin D deficiency in Hashimoto's thyroiditis during hypothyroidism: Serum vitamin D levels are lower than normal
  Interventions: Drug: Vitamin D Drops
- Patients with normal serum vitamin D during hypothyroidism in Hashimoto's thyroiditis: Serum vitamin D levels are within normal limits

INTERVENTIONS:
Drug: Vitamin D Drops — Supplement 2000IU of vitamin D, no matter the brand or manufacturer for 1 month.
  Other Names: Vitamin D
  Groups: Serum vitamin D deficiency in Hashimoto's thyroiditis during hypothyroidism

SUMMARY:
The purpose of this study is to explore the relationship between vitamin D and Hashimoto's thyroiditis and to explore whether vitamin D can play an adjuvant role in the treatment of Hashimoto's thyroiditis. Epidemiological surveys show that vitamin D deficiency rates are as high as 50%-90% in HT patients. Dietary supplementation with vitamin D has been evaluated as a way to protect the thyroid gland from autoimmune damage, but the results of randomized clinical trials are unclear.

DETAILED DESCRIPTION:
Hashimoto's thyroiditis (HT), also known as chronic lymphocytic or autoimmune thyroiditis (AITD), is a type of chronic autoimmune thyroid disease that is associated with varying degrees of hypothyroidism, thyroid autoantibody production, and lymphocytic infiltration. In China, the incidence rate showed a rising trend year by year. For the majority of HT hypothyroidism patients, synthetic levothyroxine (LT4) (first crystallized by Kendall in 1915, commercialized in the 1930s, and mass-produced in the 1960s) remains the only effective drug for HT patients. The treatment works for most patients, but is still controversial. Dietary vitamin D supplementation has been evaluated as a way to protect the thyroid from autoimmune damage, but results from randomized clinical trials have been inconclusive. Clinical studies have shown that vitamin D3 supplementation has a unique advantage in reducing TPO antibody titers. In 2014, AACE (American Association of Clinical Endocrinologists) guidelines indicated that vitamin D can be used as a complementary treatment for Hashimoto's thyroiditis. The prevalence of vitamin D deficiency in HT patients is as high as 50%-90%. Studies have shown that VD is widely used in vivo. VD can be used as an immune factor to participate in the process of immune regulation. Cells of the immune system (B cells, T cells and antigen presenting cells) can synthesize active metabolites of vitamin D due to the expression of 1α-hydroxylase (CYP27B1), which shows immunomodulatory properties. In addition, studies have shown that Vitamin D receptor (VDR) is found not only in bone, kidneys, and intestine, but also in the immune system (T and B cells, macrophages, and monocytes), reproductive system, endocrine system, muscle, brain, skin, and liver. The expression of the vitamin D receptor in these cells suggests a local role for vitamin D in immune responses. Existing genetic studies have found that most VDR can be restricted by CYP1α and vitamin D binding proteins, showing the relationship between VDR, DBP and CYP1α gene polymorphisms and thyroid autoimmune system, which affect T and B lymphocytes, dendritic cells and macrophages, as well as enzymes with CYP1α and VDR. Therefore, Vitamin D is thought to be an immune modulator.

Clinical studies have confirmed that vitamin D deficiency is more common in patients with autoimmune thyroid disease (AITD), both in children and the elderly, and in both low and high latitudes. Combining vitamin D with anti-thyroid drugs or thyroid hormones can help treat AITD by suppressing autoimmune responses and lowering serum levels of thyroid autoantibodies. However, studies have shown that vitamin D deficiency is not associated with AITD, especially early AITD. However, a study based on Asian Indian communities found only a weak inverse association between serum 25-hydroxyvitamin D values and TPO antibody titers. A 2015 meta-analysis demonstrated that vitamin D deficiency is prevalent in AITD subjects and that these subjects have low serum 25-hydroxyvitamin D levels, suggesting that lower serum 25-hydroxyvitamin D is associated with AITD disease.

There is a complex relationship between HT and serum 25-hydroxyvitamin D. It is not clear whether the decreased serum 25-hydroxyvitamin D level is one of the causes of HT hypothyroidism or a consequence of HT.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the diagnostic criteria of Hashimoto's thyroiditis in Western medicine (according to the Chinese Guidelines for the Diagnosis and Treatment of Thyroid Diseases - Thyroiditis and the Guidelines for the Diagnosis and Treatment of hypothyroidism in adults).
* Signing informed consent.

Exclusion Criteria:

* Patients with thyroid cancer;
* Other thyroid related diseases, such as Graves' disease;
* History of thyroid surgery or radioiodine therapy;
* Life history of iodine deficiency area with goiter;
* Immunosuppressive agents or immunomodulatory agents (mannan peptide, ubenamex, cyclophosphamide, incense) should be used within 1 month Polysaccharide, interferon, glucocorticoid, etc.); Other proprietary Chinese medicine (Bailing capsule, Prunella capsule, etc.)
* Patients taking chronic medications that may interfere with thyroid hormone or vitamin D metabolism;
* pregnancy plan during pregnancy or within six months;
* Severe liver and renal dysfunction;
* Serious systemic diseases, such as heart failure, stroke, and malignant tumors;
* With other autoimmune diseases: type 1 diabetes mellitus, systemic lupus erythematosus, rheumatoid arthritis, Vitiligo, autoimmune adrenal dysfunction;
* Those who are supplementing other trace elements;
* People allergic to vitamin D;
* Patients with hypercalcemia or other related diseases or mental disorders are unwilling to cooperate.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Hashimoto's thyroiditis patients with hypothyroidism.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
TPOAB in IU/ml | Data for each participant will be collected within 3 days
  Thyroid peroxisomes, a thyroid autoantibodies

SECONDARY OUTCOMES:
TGAB in IU/ml | Data for each participant will be collected within 3 days
  Thyroglobulin antibody, a thyroid autoantibody
FT3 in pmol/L | Data for each participant will be collected within 3 days
  Serum free triiodothyronine (FT3), one of the indicators reflecting thyroid function
FT4 in pmol/L | Data for each participant will be collected within 3 days
  Serum free thyroxine (FT4), one of the indicators reflecting thyroid function
TSH in uIU/ml | Data for each participant will be collected within 3 days
  Thyroid-stimulating hormone (TSH) is a hormone secreted by adenohypophysis that promotes the growth and function of thyroid gland and promotes the proliferation of thyroid follicular epithelial cells and the synthesis and release of thyroid hormone.

CONTACTS AND LOCATIONS:
Overall Officials: Yuying Cui, Study Chair — Qianfoshan Hospital